CLINICAL TRIAL: NCT01317732
Title: Calibration and Validation of MOTIONPOD(TM) for Physical Activity Evaluation in Free-living Adults
Brief Title: MOTIONPOD (TM) Validation and Calibration Study
Acronym: MOTIONPOD(TM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2010.617
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2014-03

CONDITIONS: Energy Expenditure
Keywords: Energy expenditure, physical activity, accelerometer, magnetometer, monitoring
MeSH Terms: conditions — Motor Activity | interventions — Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MOTIONPOD (TM) (Experimental)
  Interventions: Device: MOTIONPOD (TM) measures

INTERVENTIONS:
Device: MOTIONPOD (TM) measures — It is a study with a single arm. The MOTIONPOD TM measures are compared with simultaneous estimations obtained with the criteria measure (indirect calorimeter) and with existing activity monitors (heart rate monitor POLAR; different accelerometers - rT3 et Actigraph GT3X-, Actiheart, Sensewear Pro2 Armband) After physical fitness evaluation, different activity monitors are set up and the subjects perform a series of standardised activity tasks of different intensities, and well as a 30-min free activity period. Physical activity energy expenditure is measured at the end of each task using a metabolic gas analyser

SUMMARY:
In this study we propose 1) to develop a new multisensor monitoring system associating a tri-axial accelerometer and a magnetometer to measure physical activity in free-living adults, 2) to perform its calibration and assess its validity in a series of activity tasks in comparison with the measure of energy expenditure by indirect calorimetry as the criterion measure, and with existing physical activity monitors (cardiofrequencemetry and accelerometers used either alone or in combination). Briefly the subjects will perform a series of standardized activity tasks of different intensities and a 30-min free physical activity period while wearing 6 MOTIONPOD(TM) and different commercial activity monitors. Physical activity energy expenditure will be measured using a metabolic gas analyser.

Data of the 30 first subjects will be used to develop new algorithms to identify the different activity tasks and to estimate the related energy expenditures. Data of the following 30 subjects will be used to validate the MotionPOD(TM) against indirect calorimetry and existing physical activity monitors

ELIGIBILITY:
Inclusion Criteria:

* Normal-weight, overweight or obesity according to body mass index
* Low,moderate or high level of physical activity as estimated by questionnaire
* No angina and/or peripheral arterial disease symptoms or medical history

Exclusion Criteria:

* Subjects with cardiac implants
* Claustrophobic subjects
* Drug use that could affect energy expenditure
* Medical history or evolving disease which are a contra-indication for moderate physical exercise

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Estimation by the MOTIONPODTM of the physical activity energy expenditure (PAEE) during a 30-min free activity period in comparison with the measure of PAEE by indirect calorimetry | 30 minutes

SECONDARY OUTCOMES:
Identification and classification of the tasks performed during a 30-min free activity period | 30 minutes
Estimation by the MOTIONPODTM of the physical activity energy expenditure during each of the tasks performed during the experiment in comparison with 1) indirect calorimetry, 2) existing commercially activity monitors | During three hours
Intensity classification by the MOTIONPODTM of the physical activity energy expenditure during each of the tasks performed during the experiment and during the 30-min free activity period. | During three hours
  Intensity classification by the MOTIONPODTM of the physical activity energy expenditure during each of the tasks performed during the experiment and during the 30-min free activity period in comparison with 1) indirect calorimetry, 2) existing commercially activity monitors

CONTACTS AND LOCATIONS:
Overall Officials: Chantal SIMON, Pr,PhD, MD, Principal Investigator — Hospices Civils de Lyon Centre de Recherche en Nutrition Humaine Rhône-Alpes (CRNH-RA)
Locations (1):
- Hospices Civils de Lyon Centre de Recherche en Nutrition Humaine Rhône-Alpes (CRNH-RA), Pierre-Bénite, France

REFERENCES:
- [Result] Bastian T, Maire A, Dugas J, Ataya A, Villars C, Gris F, Perrin E, Caritu Y, Doron M, Blanc S, Jallon P, Simon C. Automatic identification of physical activity types and sedentary behaviors from triaxial accelerometer: laboratory-based calibrations are not enough. J Appl Physiol (1985). 2015 Mar 15;118(6):716-22. doi: 10.1152/japplphysiol.01189.2013. Epub 2015 Jan 15. PMID 25593289